CLINICAL TRIAL: NCT00826046
Title: Expanded Access of Prochymal® (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) Infusion for the Treatment of Patients Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Brief Title: Prochymal® Expanded Access for Adults Who Have Failed Steroid Treatment for Acute Graft Versus Host Disease (GVHD)
Status: No longer available | Type: Expanded Access
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Other Study IDs: 276
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Graft-Versus-Host Disease
Keywords: GVHD; Prochymal; Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — remestemcel-l

INTERVENTIONS:
Drug: Prochymal® — Patients will be treated with Prochymal twice per week at a dose of 2 x 106 hMSC/kg (actual body weight) for each of 4 consecutive weeks. Infusions will be administered at least 3 days apart.
  Other Names: Ex-vivo Cultured Adult Human Mesenchymal Stem Cells

SUMMARY:
This protocol allows for the treatment of patients, male and female, between the ages of 18 years and 70 years. Patients must have failed to respond to steroid treatment for Grade C-D acute GVHD.

DETAILED DESCRIPTION:
This is a treatment protocol to provide patients who have failed steroid treatment for acute GVHD expanded access of Prochymal. It is anticipated that a maximum of 10 patients per month for a total of 120 patients per year will be treated according to this protocol.

Patients will be treated with Prochymal twice per week at a dose of 2 x 106 human mesenchymal stem cell (hMSC)/kg (actual body weight) for each of 4 consecutive weeks. Infusions will be administered at least 3 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years to 70 years of age, inclusive.
* Biopsy confirmation of GVHD is strongly recommended, to exclude patients presenting with diarrhea or abnormal liver function tests caused by infection.
* Patients must have failed to respond to steroid treatment (methylprednisolone [≥1mg/kg/day] or equivalent) for Grades C-D acute GVHD.
* Prochymal must be administered not longer than 14 days after the initiation of systemic steroid therapy for acute GVHD.
* Prochymal must be administered either before or at the same time any additional GVHD therapy is administered
* Patients must have an adequate renal function as defined by Cockcroft-Gault equation:Calculated creatinine clearance (CrCl) > 30 mL/min
* Patients who are women of childbearing potential, must be non-pregnant, not breast-feeding, and use adequate contraception. Male patients must use adequate contraception.

Exclusion Criteria:

* Patient has stage 3 or 4 liver GVHD, bilirubin >6 mg/dl.
* Patient has stage 4 GI-GVHD.
* Patient has any underlying or current medical condition that would interfere with the evaluation of the patient including uncontrolled infection, sepsis, organ failure, etc or any medical condition that has a high probability of causing death in less than 30 days.
* Patient may not receive any other investigational agent (not approved by the FDA for any indication) concurrently for the duration of the protocol.
* Patient has evidence of a pulmonary infiltrate or diffuse alveolar hemorrhage and must not be likely to require more than 2 liters of oxygen via face mask or an estimated fractional inspired oxygen concentration (FiO2) of 28% via other delivery methods in order to sustain an O2 saturation of 92% during the next 3 days.
* Patient has a known allergy to bovine or porcine products
* Patient has a medical history of a solid tumor disease.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (3):
- United States (3):
  - Indiana BMT, Beech Grove, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York